CLINICAL TRIAL: NCT04070196
Title: Rapid Point-of-care Test for Diagnosis of Peritonitis in Peritoneal Dialysis Patients
Brief Title: Point-of-care Test for Diagnosis of Peritonitis in Peritoneal Dialysis Patients
Acronym: Periplex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Mologic Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/3152
Record Dates: First submitted 2019-08-18; First posted 2019-08-28 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Peritonitis
Keywords: Peritonitis; point-of-care test; Peritoneal Dialysis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leucocyte testing (Other): The PD effluent will be sent to the laboratory for leucocyte testing for patients presented with suspected PD peritonitis.
  Interventions: Diagnostic Test: Periplex

INTERVENTIONS:
Diagnostic Test: Periplex — Periplex test strip will be used to examine the PD effluent for peritonitis, in addition to the routine leucocyte testing of PD effluent

SUMMARY:
Peritoneal dialysis (PD) is a home-based dialysis therapy and peritonitis is a serious complication in PD. A reliable point-of-care test to detect peritonitis is important for patients to self-detect peritonitis at home as delayed diagnosis and treatment of peritonitis will translate to poor outcomes in PD patients. The study aims to examine the effectiveness of Periplex®, point-of-care test, in the diagnosis of peritonitis in PD patients.

DETAILED DESCRIPTION:
A reliable point-of-care test to detect peritonitis is indeed needed for early diagnosis of peritonitis at home and seeking medical help early.

We hypothesize that Periplex® is not inferior to routine leukocyte testing of PD Fluid effluent in the diagnosis of peritonitis. The test strip is designed to detect the inflammatory markers (IL6 and MMP-8) which are usually released during peritonitis. The strip is intended to be used in the PD patients who suspected to have symptoms of peritonitis. The target population is all adult PD patients who are followed up in Singapore General Hospital and have signs and symptoms suspected of peritonitis during the study period. The test is considered positive for peritonitis if one or both test lines appear in the window of the test strip.

The test will be performed at 2-time points, one at the presentation of peritonitis and one at the completion of antibiotics for the current episode of peritonitis, to document resolution of peritonitis.

The results of the tests will be compared with the leukocyte testing of PD effluent.

ELIGIBILITY:
Inclusion Criteria:

* Adult PD patients who are followed up in Singapore General Hospital and presented with signs and symptoms suspected of peritonitis including fever, abdominal pain or cloudy effluent will be recruited for the study.

Exclusion Criteria:

* 1. PD patients who are not followed up in SGH 2. Patients with mentally challenging conditions and who are unable to provide a valid consent 3. Non-PD patients 4. PD patients who do not have signs or symptoms suspected of peritonitis

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Test positive for peritonitis | within 24 hours of presentation with signs and symptoms suspected of peritonitis in PD patients.
  Number of participants having positive test result for peritonitis

SECONDARY OUTCOMES:
resolution of peritonitis | within 2 weeks of completion of a course of antibiotics for peritonitis
  Number of participants having negative test result for peritonitis
causal organisms for peritonitis | within a week of peritonitis
  Number of participants with gram-positive organisms, gram-negative organisms, no bacterial growth or other organisms peritonitis having test result positive for peritonitis

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore